CLINICAL TRIAL: NCT05553704
Title: Clinical Study to Compare the Possible Efficacy of Metformin in Patients With Ulcerative Colitis Treated With Mesalamine
Brief Title: Metformin in Patients With Ulcerative Colitis Treated With Mesalamine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Mounir Hussein Bahgat Internal Medicine Department Mansoura University (Unknown); Maha Mohamed Maher Internal Medicine Department Mansoura University (Unknown)
Responsible Party: Principal Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3422
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): this group will take mesalamine 1 gm three times daily for 6 months
- metformin group (Active Comparator): this group will take mesalamine 1 gm three times daily plus metformin 500 mg two times daily for 6 months
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — metformin group will take mesalamine 1 gm three times daily plus metformin 500 mg two times daily
  Arms: metformin group

SUMMARY:
Ulcerative colitis (UC) is an idiopathic, chronic inflammatory disease characterized by diffused inflammation of the colon and rectum mucosa, however, the exact underlying mechanisms of UC remain poorly understood.UC is strongly dependent on cellular immune reaction and exaggerated inflammatory response due to genetic, immune and environmental factors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Both males and females will be included
* Negative pregnancy test and effective contraception

Exclusion Criteria:

* •

  * Breast feeding
  * Significant liver and kidney function abnormalities
  * Diabetic patients
  * Colorectal cancer patients
  * Patients with severe UC
  * Patients taking rectal or systemic steroids
  * Patients taking immunosuppressives or biological therapies
  * Addiction to alcohol and / or drugs
  * Known allergy to the studied medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change in partial mayo score index | 6 months
  The Partial Mayo Score index is a non-invasive clinical scale used to assess the severity of ulcerative colitis. It is a composite of sub scores from three categories, including stool frequency, rectal bleeding, and physician's global assessment, with a total score ranging from 0-9

SECONDARY OUTCOMES:
The secondary endpoint is estimated by changes in serum IL-6 and TNF-alpha | 6 months
  The secondary endpoint is estimated by changes in serum IL-6 and TNF-alpha

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Binsaleh AY, El-Haggar SM, Hegazy SK, Maher MM, Bahgat MM, Elmasry TA, Alrubia S, Alsegiani AS, Eldesoqui M, Bahaa MM. The adjunctive role of metformin in patients with mild to moderate ulcerative colitis: a randomized controlled study. Front Pharmacol. 2025 Mar 19;16:1507009. doi: 10.3389/fphar.2025.1507009. eCollection 2025. PMID 40191419
- [Derived] El-Haggar SM, Hegazy SK, Maher MM, Bahgat MM, Bahaa MM. Repurposing metformin as adjuvant therapy in patients with ulcerative colitis treated with mesalamine: A randomized controlled double-blinded study. Int Immunopharmacol. 2024 Sep 10;138:112541. doi: 10.1016/j.intimp.2024.112541. Epub 2024 Jun 24. PMID 38917525